CLINICAL TRIAL: NCT02335567
Title: Use of in Vivo 3T MR to Characterize Carotid Plaque in Patients and Correlate MR Findings With Symptoms
Acronym: 3TMR
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Kevin DeMarco, Associate Professor, Michigan State University
Other Study IDs: GE sequence
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Carotid Plaque Hemorrhage Appearance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: there is no intervention

SUMMARY:
To compare two competing newly designed 3D sequences for black blood carotid plaque imaging techniques with the industry standard 2D sequnce for black blood.

DETAILED DESCRIPTION:
To utilize a 3D sequence instead of the usual 2D commonly standard industry sequence that is supplied by the various manufacturers.

Patients with greater than 50% stenosis that are 3T compatible are imaged using the two sequences to compare which sequences better visualize the plaque and it's characteristics

The purpose is to validate the ability of the new 3D sequence to detect and measure any plaque hemorrhage as well as to identify region sof Type 1 hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 50% stenosis of the carotid arteries that are safe to undergo MRI imaging

Exclusion Criteria:

* Patients that are determined to no be safe to undergo MR imaging due to implants

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with 50% asymptomatic stenosis of the carotid artery that are safe to undergo 3 tesla MRI imaging.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Appearance of intraplaque hemorrhage | 1 day of scan
  what radiologist interperts

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University - Department of Radiology, East Lansing, Michigan, United States

REFERENCES:
- [Background] Ota H, Reeves MJ, Zhu DC, Majid A, Collar A, Yuan C, DeMarco JK. Sex differences of high-risk carotid atherosclerotic plaque with less than 50% stenosis in asymptomatic patients: an in vivo 3T MRI study. AJNR Am J Neuroradiol. 2013 May;34(5):1049-55, S1. doi: 10.3174/ajnr.A3399. Epub 2012 Nov 29. PMID 23194832
- [Background] DeMarco JK, Willinek WA, Finn JP, Huston J 3rd. Current state-of-the-art 1.5 T and 3 T extracranial carotid contrast-enhanced magnetic resonance angiography. Neuroimaging Clin N Am. 2012 May;22(2):235-57, x. doi: 10.1016/j.nic.2012.02.007. PMID 22548930
- [Background] Mughal MM, Khan MK, DeMarco JK, Majid A, Shamoun F, Abela GS. Symptomatic and asymptomatic carotid artery plaque. Expert Rev Cardiovasc Ther. 2011 Oct;9(10):1315-30. doi: 10.1586/erc.11.120. PMID 21985544
- [Background] Ota H, Reeves MJ, Zhu DC, Majid A, Collar A, Yuan C, DeMarco JK. Sex differences in patients with asymptomatic carotid atherosclerotic plaque: in vivo 3.0-T magnetic resonance study. Stroke. 2010 Aug;41(8):1630-5. doi: 10.1161/STROKEAHA.110.581306. Epub 2010 Jul 8. PMID 20616325
- [Background] Underhill HR, Hatsukami TS, Cai J, Yu W, DeMarco JK, Polissar NL, Ota H, Zhao X, Dong L, Oikawa M, Yuan C. A noninvasive imaging approach to assess plaque severity: the carotid atherosclerosis score. AJNR Am J Neuroradiol. 2010 Jun;31(6):1068-75. doi: 10.3174/ajnr.A2007. Epub 2010 Jan 21. PMID 20093315
- [Result] DeMarco JK, Huston J 3rd. Imaging of high-risk carotid artery plaques: current status and future directions. Neurosurg Focus. 2014 Jan;36(1):E1. doi: 10.3171/2013.10.FOCUS13384. PMID 24380475
- [Result] Zhu DC, Vu AT, Ota H, DeMarco JK. An optimized 3D spoiled gradient recalled echo pulse sequence for hemorrhage assessment using inversion recovery and multiple echoes (3D SHINE) for carotid plaque imaging. Magn Reson Med. 2010 Nov;64(5):1341-51. doi: 10.1002/mrm.22517. PMID 20574968
- [Result] Zhu DC, Ferguson MS, DeMarco JK. An optimized 3D inversion recovery prepared fast spoiled gradient recalled sequence for carotid plaque hemorrhage imaging at 3.0 T. Magn Reson Imaging. 2008 Dec;26(10):1360-6. doi: 10.1016/j.mri.2008.05.002. Epub 2008 Jun 25. PMID 18583079